CLINICAL TRIAL: NCT01378897
Title: A Telehealth Innovation to Support Weight Loss
Brief Title: Bariatric Surgery Telemedicine Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI decided to not initiate this study.
Sponsor: Baystate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BH-11-059
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
Keywords: bariatric surgery; gastric bypass surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MedSignals®pillbox,Omron pedometer,VitalSignals®weight scale — Participants will use three home monitoring devices (i.e., weight scale, pedometer, pillbox) for two months. In addition, participants will receive weekly phone calls from the study's bariatric dietician during weeks 1-4 of the study and then receive biweekly calls during the second month. The structured phone calls (approximately 10-15 minutes each call) will focus on discussing the patient's adherence data, discussing any barriers to adherence, and providing tailored patient education.

SUMMARY:
The purpose of this study is to evaluate a new educational program for people who have recently had gastric bypass surgery. This program involves both the use of newly developed wireless home monitoring technology (medication box, weight scale, and pedometer) and telephone-based, individually tailored health counseling with a bariatric dietician.

DETAILED DESCRIPTION:
Obesity, defined as a body mass index (BMI) >30 in kg/m2, has reached epidemic levels in the United States (US). Morbid obesity, which is classified as a BMI>=40, is the fastest growing obesity category. It has increased 52% between 2000 and 2005, to now affect 15 million US adults. Morbid obesity is associated with serious medical co-morbidities, and these obesity-related diseases have a significant impact on the individual patient, as well as on our healthcare system as a whole. Gastric bypass surgery is the only current effective treatment for MO. Approximately 220,000 operations were carried out in 2008, making it one of the most commonly performed procedures in the U.S. The most common form (80%) of bariatric surgery performed in the U.S. is laparoscopic gastric bypass (LGB). While there has been considerable clinical focus on multidisciplinary pre-surgical screening regarding medical, behavioral, and psychosocial suitability of candidates for bariatric surgery, there is a paucity of post-surgical follow-up examining behavioral adaptation and adherence. The purpose of this study is to examine such post-surgical behavioral components that are relevant to weight loss surgery. Specifically, the investigators will assess the feasibility, reliability, usability, and satisfaction of some newly developed wireless home monitoring technology (i.e., medication box, weight scale, and pedometer) in a group of patients who have recently had gastric bypass surgery. A prospective cohort study design will be conducted. Questionnaire data will be collected and data analysis will be descriptive in nature.

ELIGIBILITY:
Inclusion Criteria:

* 6 weeks-1 year post gastric bypass surgery
* > 18 years of age
* English-speaking and able to read and understand consent form and study questionnaires.
* Land line analog telephone service at home

Exclusion Criteria:

* Suffered unexpected complications from surgery as judged by the surgeons
* Anyone judged not fit to participate in the study, as per the surgeon or dietician's clinical judgment
* Weight >440 lbs. at enrollment (upper limit of our weight scale)
* Planning to relocate from the area within the next 2-3 months (i.e., during study timeframe)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
usability questionnaire | 2 month
  This pilot study involves the collection of descriptive data to assess feasibility, usability, and satisfaction with the devices. ). The method for collecting study data will be questionnaires (i.e., usability questionnaire, treatment satisfaction questionnaire, and feasibility questionnaire) and electronic data from the device downloads.

CONTACTS AND LOCATIONS:
Overall Officials: Garry W Welch, PhD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States